CLINICAL TRIAL: NCT07298447
Title: An Open-Label Study of Donidalorsen in Pediatric Patients Age 2 to Less Than 12 Years Old With Hereditary Angioedema
Brief Title: Donidalorsen Treatment in Children With Hereditary Angioedema
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 721744-CS8; U1111-1326-8613 (Other: WHO Universal Trial Number (UTN)); 2025-523499-22-00 (Other: EU Trial No.)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — donidalorsen; IONIS-PKK-LRx

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Donidalorsen: Group 1 (Experimental): Participant weighing 9 kilograms (kg) to less than (<)26 kg, will be administered donidalorsen over the period of one year.
  Interventions: Drug: Donidalorsen
- Donidalorsen: Group 2 (Experimental): Participant weighing greater than or equal to (≥)26 kg to <41 kg, will be administered donidalorsen over the period of one year.
  Interventions: Drug: Donidalorsen
- Donidalorsen: Group 3 (Experimental): Participant weighing ≥41kg, will receive donidalorsen over the period of one year.
  Interventions: Drug: Donidalorsen

INTERVENTIONS:
Drug: Donidalorsen — Donidalorsen will be administered by subcutaneous (SC) injection.
  Other Names: ISIS 721744; IONIS-PKK-LRx

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of donidalorsen in pediatric participants with hereditary angioedema (HAE) Type I (HAE-1) or Type II (HAE-2).

DETAILED DESCRIPTION:
This is an open-label study to evaluate the safety, efficacy, and pharmacokinetics (PK) and pharmacodynamics (PD) of donidalorsen in pediatric participants age 2 to less than 12 years old with HAE Type I (HAE-1) or Type II (HAE-2). The study consists of 3 parts: 1) a 3-month Screening Period, 2) a one-year Treatment Period, and 3) a 3-month Post-Treatment Period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must be between the ages of 2 and less than 12 years, inclusive, at the time of informed consent and, as applicable, assent.
2. Must weigh at least 9 kg at the time of informed consent and, as applicable, assent.
3. Documented diagnosis of HAE-1/HAE-2 based upon both of the following:

   1. Documented clinical history consistent with HAE (SC or mucosal, non-pruritic swelling episodes without accompanying urticaria).
   2. Diagnostic testing results that confirm HAE-1/HAE-2: C1-inhibitor (C1-INH) functional level <50% normal level AND complement factor C4 level below the lower limit of normal (LLN); OR a known pathogenic mutation in the SERPING1 gene.

Key Exclusion Criteria:

1. Must not have any screening laboratory abnormalities or any other clinically significant abnormalities during screening that would render a participant unsuitable for inclusion.
2. Must not have been treated with another investigational drug, biological agent, or device within 1 month of Screening, or 5 half-lives of investigational agent, whichever is longer.
3. Concurrent diagnosis of any other type of recurrent angioedema, including idiopathic angioedema or HAE with normal C1-INH (HAE-nC1-INH or Type III).

Note: Other protocol-specified inclusion/exclusion criteria may apply.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | over the period of approximately 17 months
Maximum Plasma Concentration (Cmax) of Donidalorsen | over the period of approximately 17 months
Maximum Time to Reach Cmax (Tmax) of Donidalorsen | over the period of approximately 17 months
Trough Plasma Concentration (Ctrough) of Donidalorsen | over the period of approximately 17 months

SECONDARY OUTCOMES:
Time-Normalized Number of Investigator-Confirmed HAE Attacks (per Month) | over the period of 12 months
Percentage of Investigator-Confirmed HAE Attack-free Participants | over the period of 12 months
Time-Normalized Number of Moderate or Severe Investigator-Confirmed HAE Attacks (per Month) | over the period of 12 months
Number of Participants with a Clinical Response Defined as a ≥ 50 Percent (%), ≥ 70% and ≥ 90% Reduction from Baseline in Investigator-Confirmed HAE Attack Rate | over the period of 12 months
Time-Normalized Number of Investigator-Confirmed HAE Attacks Requiring Rescue Treatment | over the period of 12 months
Change From Baseline in Prekallikrein (PKK) Levels in Plasma | over the period of 12 months
Percent Change From Baseline in PKK Levels in Plasma | over the period of 12 months
Changes in Pediatrics Quality of Life (PedsQL) Scores for Participants | over the period of 12 months

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/